CLINICAL TRIAL: NCT07373912
Title: Impact of Adding Instrument-assisted Soft Tissue Mobilization to Mulligan Therapy in Patients With Cervicogenic Headache
Acronym: CGH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Youssef Ahmed Mahmoud, principle investigator : doaa youssef ahmed mahmoud, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006193
Record Dates: First submitted 2026-01-21; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cervicogenic Headache
Keywords: Instrument Assisted Soft Tissue Mobilization; mulligan therapy
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: instrument-assisted soft tissue mobilization, Mulligan therapy, and postural correction exercises
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- instrumeted assissted soft tissue mobilization and mulligan therapy (Experimental): twenty patients will receive IASTM, mulligan therapy and postural correction exercises three times per week for 6 weeks.
  Interventions: Other: instrumeted assissted soft tissue mobilization and mulligan therapy; Other: mulligan therapy; Other: postural correction exercises
- mulligan therapy (Experimental): Twenty patients will receive Mulligan therapy and postural correction exercises three times per week for 6 weeks.
  Interventions: Other: mulligan therapy; Other: postural correction exercises
- postural correction exercises (Active Comparator): Twenty patients will receive postural correction exercises three times per week for 6 weeks.
  Interventions: Other: postural correction exercises

INTERVENTIONS:
Other: instrumeted assissted soft tissue mobilization and mulligan therapy — the patients will receive IASTM tools over the length of targeted muscles (descending fiber of trapezius, suboccipitalis muscles ) for 5 minutes. also, SNAG technique; Each patient will be asked to sit comfortably, and the treating therapist will stand beside the patient. The patient's head will be free and cradled between the therapist's right forearm and body, and the therapist stand at the patient's right side. The therapist then will place his right index, middle, and ring fingers at the base of the occiput and kept his right little finger over the spinous process of C2. Next, with the lateral border of his left thenar eminence, gentle pressure will be applied in a ventral and upward direction(45 degrees) over the right little finger. finally postural correction execises
  Arms: instrumeted assissted soft tissue mobilization and mulligan therapy
Other: mulligan therapy — SNAG technique; Each patient will be asked to sit comfortably, and the treating therapist will stand beside the patient. The patient's head will be free and cradled between the therapist's right forearm and body, and the therapist stand at the patient's right side. The therapist then will place his right index, middle, and ring fingers at the base of the occiput and kept his right little finger over the spinous process of C2. Next, with the lateral border of his left thenar eminence, gentle pressure will be applied in a ventral and upward direction(45 degrees) over the right little finger. Finally, postural correction exercises will be addedd
  Arms: instrumeted assissted soft tissue mobilization and mulligan therapy; mulligan therapy
Other: postural correction exercises — the exercises will incluse, Stretching exercises for the sternocleidomastoids,the Scalenes,upper fibers of trapezius and strengthening exercises for cervical muscles

SUMMARY:
this study will be conducted to investigate the impact of adding Instrument assisted soft tissue mobilization technique to mulligan therapy in patients with cervicogenic headache

DETAILED DESCRIPTION:
Cervicogenic headache (CGH) has seen a notable rise in prevalence in recent years, substantially impairing patients' daily functioning and occupational productivity. Despite its considerable burden, CGH remains frequently underdiagnosed and inadequately managed, often progressing to a chronic state that heightens the risk of work absenteeism and long-term disability and as the most common type of pain disorders, affecting 66% of the global population, represent a major public health concern due to their detrimental impact on quality of life and economic productivity . Epidemiological data indicate that CGH affects 4.1% of the general population, with prevalence escalating to 17.5% among individuals with severe headaches.Instrument Assisted Soft Tissue Mobilization using Graston (GT®) tool is regarded as one the most advanced and promising methods ,utilizing a specially designed instrument to adress a variety of soft tissue pathologies such as myofascial adhesions , scar tissue restriction , tissue thickenings, ridges, fibrotic nodules, crystalline deposits . this technique works by generating a mobilizing effect ,which contributes to pain reduction ,enhanced range of motion and improved overall function.The Mulligan manual technique is considered one of the most effective forms of manipulations. In contrast to conventional mobilization, which depends entirely on the therapist, Mulligan proposed that applying pressure to the spinous processes while the patient is in a weight-bearing position would cause the facet joints to glide in a coordinated ,parallel direction . simultaneously ,this approach involve the patient's active participation during movemwnt in order to achieve the perfect therapeutic outcomes

ELIGIBILITY:
Inclusion Criteria:

-Unilateral CGH presentation

* Age group above 18 years' old
* History of chronic CGH (>3 months)
* CGH owing to cervical spine (neck) dysfunction
* Reduced cervical motion
* Neck stiffness and movement restriction

Exclusion Criteria:

* Participants with other types of headache (migraine headache)
* Headache owing to other causes (sinus, tumor, neural, and tempero-mandibular joint issues)
* Any contraindications to manual and manipulative therapy (fracture, instability, osteoporosis and neural symptoms)
* Taking analgesics or corticosteroids and migraine-specific medications, such as triptans
* Metastasis
* Cardiac conditions (stroke and syncope)
* Neurological conditions (radiculopathy, myelopathy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
neck disability | up to 6 weeks
  Assessment of neck function was performed by Arabic neck disability index. It is a valid and reliable tool in the assessment of neck function. It contains ten category/classes. Each category contains six choices (zero-five).Score from zero to four no disability, from five to 15 this is mild, From 15 to 24 this is moderate, from 25 to 34 this is severe, more than 34 this is a complete disability

SECONDARY OUTCOMES:
pain intensity | up to 6 weeks
  The scale will be used is the VAS, which consists of a line, usually 10 cm long, ranging from no pain or discomfort (zero) , to the worst pain that could possibly feel (10)
cervical range of motion | up to six weeks
  The CROM device will be used to assess cervical range of motion. it is headmounted equipment consists of a plastic frame placed on the head over the nose and the ears, secured by a Velcro strap. Two independent inclinometers, 1 in the sagittal plane and 1 in the frontal plane, are attached to the frame and indicate the position of the head with respect to the line of gravity. A third inclinometer is positioned in the horizontal plane and indicates the position of the head in rotation, with respect to a reference position
muscle stiffness | up to six weeks
  The MyotonPRO (Myoton AS, Tallinn, Estonia) is a recently introduced device that can objectively measure the mechanical properties of muscles including analyzing muccsle stiffness (N/m).
  The measurement procedure involved pressing the device against the skin, with a force of 0.18 N and instantly applying an impulse of 0.4 N for duration of 15 ms. The skin surface oscillation induced by the\ MyotonPRO was measured
headache frequency | up to six weeks
  the number of days the subjects experienced headaches (frequency)
headache duration | up to six weeks
  the total number of hours they experienced headaches (duration)
medication intake | up to 6 weeks
  The frequency with which they used painkillers (medication intake) for their headaches were also noted